CLINICAL TRIAL: NCT06627348
Title: Hilotherapy for Prevention of Chemotherapy-induced Peripheral Polyneuropathy - a Unicentric, Prospective-controlled, Randomized Clinical Trial for Comparison of Local Hilotherapy Vs. No Therapy to Prevent Peripheral Polyneuropathy During Taxan-based Chemotherapy Regimen
Brief Title: Hilotherapy for Prevention of Chemotherapy-induced Peripheral Polyneuropathy
Acronym: HiPPo
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ulm (Other)
Collaborators: Hilotherm (Unknown)
Responsible Party: Principal Investigator, Prof. Wolfgang Janni, Director of the Department of Gynecology and Obstetrics, University of Ulm
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HIPPO
Record Dates: First submitted 2023-10-20; First posted 2024-10-04 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Equipment and Supplies
Keywords: Chemo-induced Peripheral Polyneuropathy; Taxan; Hilotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hilotherapy (Active Comparator): Cooling of hands and feet during Taxan-based chemotherapy
  Interventions: Device: Hilotherm ChemoCare
- No Cooling (No Intervention): No cooling of hands and feet during Taxan-based chemotherapy

INTERVENTIONS:
Device: Hilotherm ChemoCare — Hilotherapy
  Arms: Hilotherapy

SUMMARY:
Prospective study of hilotherapy of hands and feet as prevention of chemotherapy-induced peripheral polyneuropathy induced by Taxan-based chemotherapy regimen that are used in the therapy of breast cancer and genital malignoma of the women.

DETAILED DESCRIPTION:
In this trial, patients receiving Taxan-based chemotherapy regimen e.g. paclitaxel, nab-paclitaxel or docetaxel in gynecological malignancies such as ovarian cnacer, breast cancer, endometrial cancer or cervical cancer will either receive cooling of hands and feet during the application of above-mentioned substances or not. The cooling will be provided by a machine called Hilotherm ChemoCare unit and will be administered constantly at a temperature of 15-17°C. Randomization will be 50:50.

if a patient is randomized in the non-interventional arm, no cooling is allowed during the application of the chemotherapy.

To assess the occurance and the extent of peripheral neuropathy, a neurological examination will take place before the start of chemotherapy, in the middle of the planned cycles of chemotherapy and after the completion of the regimen.

Quality of life and the subjective impacts of peripheral neuropathy will be evaluated via questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Written consent for participation in this trail
* Age ≥18 years
* Female
* Breast or genital cancer of the woman
* Planned application of a Taxan-based chemotherapy regimen (Paclitaxel, Nab-Paclitaxel, Docetaxel) independent of the therapy line
* Taxan- and Platin-naivity
* Sufficient knowledge of the German language to assure an adequat survey of patient's history

Exclusion Criteria:

* pre-existing peripheral polyneuropathy
* chemotherapy with taxan- and/or carboplatin-based regimens in a preceding therapy
* Existence of one of the following diseases: Diabetes mellitus (of any type), neurological diseases that are involving peripheral nerve damage (e.g. Multiple Sclerosis, Amytrophic lateral sclerosis, Parkinson's disease), chronic pain syndrome, Cryoglobulinemia, cold hemagglutination, cold hives / cold contact hives, Raynaud's disease, significant peripheral artery disease,
* Lack of knowledge of German
* Males

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-04-17 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
incidence of peripheral polyneuropathy | Up to one year after the end of chemotherapy.
  The primary endpoint of this study is the comparison of the incidence of a peripheral polyneuropathy (clinical Total Neuropathy Score cTNS ≥ 11) in patients with gynecologic malignoma that are undergoing Taxan-based chemotherapy regimen with or without a preventive hilotherapy of hands and feet.

SECONDARY OUTCOMES:
Changes in the result of electrophysical examinations | From the beginning to the end of chemotherapy, exact time frame depending on the chemotherapy regimen, assessed up to 30 weeks.
  Changes in the result of electrophysical examinations before and after chemotherapy.
Adverse effects of hilotherapy | Up to one year after the end of chemotherapy.
  Adverse effects of hilotherapy documented as any adverse event.
Tolerance of chemotherapy | From the beginning to the end of chemotherapy, exact time frame depending on the chemotherapy regimen, assessed up to 30 weeks.
  Tolerance of chemotherapy measured as the proportion of patient with dose reduction or premature end of chemotherapy.
Patient reported Quality of Life | Up to one year after the end of chemotherapy.
  Quality of Life of patients measured with the EORTC QLQ-C30 questionnaire
Residual Symptoms of Chemotherapy-induced polyneuropathy | Up to one year after the end of chemotherapy.
  Comparison of the time of regression, cTNS score of persisting symptoms and amount of patients without residues after end of chemotherapy and follow-up between patients with and without preventive hilotherapy.
Subjective extent of CIPN | Up to one year after the end of chemotherapy.
  Subjective extent of CIPN as measured with the EORTC QLQ-CIPN20 (quality of life questionnaire regarding chemotherapy-induced peripheral neuropathy with 20 questins) questionnaire.
  The qustionnaire consits of 20 items on 3 scales. The minimum is 0, the maximum is 100 points. The higher the score, the worse the CIPN.
Acceptance of hilotherapy | From the beginning to the end of chemotherapy, exact time frame depending on the chemotherapy regimen, assessed up to 30 weeks.
  Acceptance of hilotherapy measured as the amount of patients that have to stop local cold application during a session (up to 5 minutes) or terminate earlier or stop the treament completely for the rest of chemotherapy.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Ulm, Ulm, Baden-Wurttemberg, Germany